CLINICAL TRIAL: NCT05572320
Title: Platelet Function and Neurological Events Following Carotid Thromboendarterectomy
Brief Title: Platelet Function and Neurological Events
Acronym: MULTINEUR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Fabrizio Monaco, Head of Cardiothoracic and Vascular Anesthesia, Scientific Institute San Raffaele
Other Study IDs: CE:83/INT/2022
Record Dates: First submitted 2022-09-15; First posted 2022-10-07 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute; Carotid Artery Diseases
Keywords: Carotid thromboendarterectomy; Thromboembolic Stroke; Platelet function; Aggregometry; Vascular surgery; mortality; neurological events
MeSH Terms: conditions — Stroke; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Platelet Aggregometry Testing — 1.6 ml of blood collected in hirudin-coated tubes before the surgery
  Other Names: Multiple Electrode Aggregometry (Multiplate) device

SUMMARY:
Several studies have shown an association between platelet function and stroke in patients undergoing carotid thromboendarterectomy (TEA).

The present study will assess the correlation between platelet function evaluated by the impedance aggregometry and neurological events in patients undergoing carotid TEA.

DETAILED DESCRIPTION:
Carotid thrombendarterectomy (TEA) is effective in preventing strokes which are a major cause of mortality and morbidity. Nevertheless, almost 10% of patients undergoing TEA develop a transient and/or permanent neurological injury. There is a growing body of evidence that platelet function is associated with perioperative neurological events in this setting, although the vast majority of patients undergoing carotid TEA are already on antiplatelet agents. The aim of the present study will be to assess the correlation between the platelet function evaluated by the impedance aggregometry (Multiplate ® Analyzer, Roche, Basel, Switzerland) and neurological events in patients undergoing carotid TEA.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Carotid Artery Diseases undergoing carotid thrombendarterectomy
* Signed consent

Exclusion Criteria:

* Atrial fibrillation
* New oral anticoagulant
* Oral Vitamin k inhibitors
* Platelet count <80000 per microliter
* Ongoing ischemic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing carotid thromboendoarterectomy
Sampling Method: Probability Sample
Enrollment: 386 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Platelet function and neurological events | immediately before the surgery
  The platelet function will be evaluated by Multiple Electrode Aggregometry (Multiplate). It will be asses the correlation between thrombin receptor activator peptide 6 (TRAP test), adenosine-5'-diphosphate (ADP test) and arachidonic acid (ASPI test) expressed in arbitrary units area under the curve and neurological events in patients undergoing carotid thrombendarterectomy
TRAP, ADP and ASPI thresholds to predict neurological events | immediately before the surgery
  It will be find the best cut-off for TRAP, ADP and, ASPI in predicting neurological events

SECONDARY OUTCOMES:
Occurence of thromboembolic neurological events | within 1 month of patients' enrolled or before the hospital discharge
Occurrence of any complications | within 1 month of patients' enrolled or before the hospital discharge
  Occurrence of surgical and medical complications
6 months and 1 year mortality | 6 months and 1 year
  Mortality at 6 months and 1 years after carotid surgery
6 months and 1 year neurological events | 6 months and 1 year
  Occurrence of neurological events after 6 months and 1 year after the procedure

OTHER OUTCOMES:
Assesment of the health state at 6 months and 1 year after surgery | 6 months and 1 year
  The health state will be evaluated by EuroQol 5-dimensions 3 level test at 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Monaco, MD, Principal Investigator — San Raffaele Scientific Institute
Locations (1):
- Scientific Institute San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ball STE, Taylor R, McCollum CN. Resistance to Antiplatelet Therapy Is Associated With Symptoms of Cerebral Ischemia in Carotid Artery Disease. Vasc Endovascular Surg. 2020 Nov;54(8):712-717. doi: 10.1177/1538574420947235. Epub 2020 Aug 28. PMID 32856558
- [Background] Reavey-Cantwell JF, Fox WC, Reichwage BD, Fautheree GL, Velat GJ, Whiting JH, Chi YY, Hoh BL. Factors associated with aspirin resistance in patients premedicated with aspirin and clopidogrel for endovascular neurosurgery. Neurosurgery. 2009 May;64(5):890-5; discussion 895-6. doi: 10.1227/01.NEU.0000341904.39691.2F. PMID 19287328
- [Background] Sacco S, Stracci F, Cerone D, Ricci S, Carolei A. Epidemiology of stroke in Italy. Int J Stroke. 2011 Jun;6(3):219-27. doi: 10.1111/j.1747-4949.2011.00594.x. PMID 21557809